CLINICAL TRIAL: NCT01351077
Title: A Study to Determine if CHICA Can Improve Developmental Screening
Brief Title: The CHICA Developmental Screening Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Aaron Carroll, Assoc. Prof of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHICA_DevScreen_Study; R01HS017939 (AHRQ)
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-04

CONDITIONS: Developmental Delay
Keywords: Developmental Delay
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHICA DevScreen Module (Experimental): This arm will get the CHICA Developmental Screening Module
  Interventions: Other: CHICA DevScreen Module
- CHICA DevScreen Control (No Intervention): This arm will get CHICA without the developmental screening module

INTERVENTIONS:
Other: CHICA DevScreen Module — This module assists in the diagnosis and management of developmental screening
  Arms: CHICA DevScreen Module

SUMMARY:
The aims of this study are to (1) Expand and modify an existing computer-based decision support system (CHICA) to include the 2006 AAP developmental surveillance and screening algorithm; (2) Evaluate the effect of the CHICA system on the developmental surveillance and screening practices of four pediatric clinics; (3) Evaluate the effect of the CHICA system on referrals for developmental and medical evaluations as well as early developmental intervention/early childhood services for those children identified as having concerning developmental screening results; and (4) Develop a cohort of children with identified developmental disabilities that can be followed over time in order to look at the end results/effects of developmental screening

DETAILED DESCRIPTION:
Between 12 and 16% of children in the United States have a developmental disability. Research has demonstrated that early intervention programs are not only essential for improved outcomes in these children, but also cost-effective. As a result, there has been a push within the pediatric medical community to identify children with developmental delays or disabilities as early as possible. Currently, most pediatric primary care providers do not use standardized methods for developmental surveillance and screening. Instead they rely on intuition and clinical judgment which has been shown to have limitations when compared with standardized screening methods. Researchers and physician organizations such as the AAP have called on pediatric primary care providers to institute a standardized approach for the identification of developmental delays that includes both developmental surveillance and screening. In fact, the AAP recently published an algorithm for developmental surveillance and screening within a primary care setting. Physicians, however, cite several barriers to the implementation of these recommendations within their practices, including lack of time, lack of office staff, inadequate reimbursement, and language barriers.

The investigators have developed a novel computer decision support system (CDSS) for implementing clinical guidelines and algorithms within pediatric practices called CHICA. The investigators believe that this CDSS has the potential to address the barriers cited in previous studies as obstacles specific to the implementation of developmental surveillance and screening within primary care practices. CDSS will allow for developmental surveillance and screening to fit within the workflow of a busy pediatric practice without requiring an additional investment of time on the part of the physician and without requiring additional office staff.

The aims of this study are to (1) Expand and modify an existing computer-based decision support system (CHICA) to include the 2006 AAP developmental surveillance and screening algorithm; (2) Evaluate the effect of the CHICA system on the developmental surveillance and screening practices of four pediatric clinics; (3) Evaluate the effect of the CHICA system on referrals for developmental and medical evaluations as well as early developmental intervention/early childhood services for those children identified as having concerning developmental screening results; and (4) Develop a cohort of children with identified developmental disabilities that can be followed over time in order to look at the end results/effects of developmental screening

ELIGIBILITY:
Inclusion Criteria:

* This study will involve the analysis of data collected in the care of children seen in four IUMG-PC pediatric clinics. For aim 2 of the study all children between the ages of 0 and 3 seen in the four study clinics will be eligible for and will be participants in the study.

For aim 3 of the study, a child is eligible for participation if they are younger than 5 years of age, have a concerning developmental screening result, and are seen in one of the four clinics participating in this study. Additionally, these children cannot have a previous diagnosis of a developmental disorder and at least one of the child's parents must speak English.

Exclusion Criteria:

* For aim 3, having no parents who can speak English

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron E Carroll, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Children's Health Services Research, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carroll AE, Bauer NS, Dugan TM, Anand V, Saha C, Downs SM. Use of a computerized decision aid for developmental surveillance and screening: a randomized clinical trial. JAMA Pediatr. 2014 Sep;168(9):815-21. doi: 10.1001/jamapediatrics.2014.464. PMID 25022724

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CHICA DevScreen Module | CHICA DevScreen Control
Started | 180 | 180
Completed | 180 | 180
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHICA DevScreen Module | CHICA DevScreen Control | Total
Number analyzed (Participants) | 180 | 180 | 360
Age, Continuous [Mean (Standard Deviation); unit: months] | 19.8 (5.1) | 23.7 (6.5) | 21.8 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 91 | 188
  Male | 83 | 89 | 172
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 51 | 164 | 215
  Hispanic | 117 | 11 | 128
  White/Asian | 11 | 4 | 15
  Other | 1 | 1 | 2
Insurance [Count of Participants; unit: Participants]
  Advantage/Commercial | 8 | 6 | 14
  Self-pay | 12 | 2 | 14
  Medicaid | 160 | 171 | 331

OUTCOME MEASURES:

1. Primary Outcome: Number of Children Screened for Developmental Delay
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | CHICA DevScreen Module | CHICA DevScreen Control
Number analyzed (Participants) | 180 | 180
Participants | 153 | 44

2. Secondary Outcome: Age of Children Diagnosed With Developmental Delay
Time Frame: one year
Population: The denominator was only children diagnosed with developmental delay
Measure: Mean (Standard Deviation); unit: months
Arm/Group | CHICA DevScreen Module | CHICA DevScreen Control
Number analyzed (Participants) | 19 | 12
months | 19.8 (5.1) | 23.8 (6.5)

3. Other Pre Specified Outcome: Number of Children With a Positive Screen
Time Frame: one year
Population: The denominator was number of children for whom a standard developmental screening tool was administered
Measure: Count of Participants; unit: Participants
Arm/Group | CHICA DevScreen Module | CHICA DevScreen Control
Number analyzed (Participants) | 153 | 44
Participants | 30 | 8

4. Other Pre Specified Outcome: Number of Children Referred for Evaluation and Services When There Was a Positive Screening Result
Time Frame: one year
Population: The denominator was the number of children with a positive screen
Measure: Count of Participants; unit: Participants
Arm/Group | CHICA DevScreen Module | CHICA DevScreen Control
Number analyzed (Participants) | 30 | 8
Participants | 22 | 4

5. Other Pre Specified Outcome: Number of Patients Whose Referred Evaluations and Services Were Completed
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | CHICA DevScreen Module | CHICA DevScreen Control
Number analyzed (Participants) | 22 | 4
Participants | 12 | 1

ADVERSE EVENTS:
Time Frame: two years
Arm/Group | CHICA DevScreen Module | CHICA DevScreen Control
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/180
Other Adverse Events (participants affected / at risk) | 0/180 | 0/180

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No